CLINICAL TRIAL: NCT00692978
Title: The Pharmacokinetics of Inhaled Fluticasone Propionate Delivered as Monodisperse Aerosols
Brief Title: Pharmacokinetics of Inhaled Monodisperse Fluticasone Propionate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 08/H0712/63
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Healthy; Asthma
Keywords: Monodisperse aerosols; Healthy Volunteers; Asthmatics; Pharmacokinetics; Randomized
MeSH Terms: conditions — Asthma | interventions — Metered Dose Inhalers

STUDY DESIGN:
Intervention Model Description: Two groups (asthma and healthy) go through different particle size of monodisperse aerosol treatments
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma (Experimental): Asthma patients
  Interventions: Drug: Fluticasone Propionate_1.5; Drug: Fluticasone Propionate_3; Drug: Fluticasone Propionate_6; Drug: FP From Active 250 ug MDI Inhaler
- Healthy volunters (Active Comparator): Healthy participants
  Interventions: Drug: Fluticasone Propionate_1.5; Drug: Fluticasone Propionate_3; Drug: Fluticasone Propionate_6; Drug: FP From Active 250 ug MDI Inhaler

INTERVENTIONS:
Drug: Fluticasone Propionate_1.5 — Dose 50 micrograms (total dose), Monodisperse aerosol with particle size of drug 1.5 micros, inhaled
Drug: Fluticasone Propionate_3 — Dose 50 micrograms (total dose), Monodisperse aerosol with particle size of drug 3.0 microns, inhaled
Drug: Fluticasone Propionate_6 — Dose 50 micrograms (total dose), Monodisperse aerosol with particle size of drug 6.0 microns, inhaled
Drug: FP From Active 250 ug MDI Inhaler — Monodisperse aerosols inhaled of Fluticasone Propionate at 250micrograms dose with active MDI inhaler

SUMMARY:
Asthma is most effectively treated by delivering inhaled drugs from an inhaler (puffer) directly into the lungs. Inhaled steroids are used in asthmatic patients to dampen down lung inflammation, which unchecked, can often lead to patient symptoms. Inhalers deliver a mist containing particles of lots of different sizes (like hairsprays). Medical puffers used by patients produce a 'coarse' mist of drug particles, which have the potential for side effects, as different sized particles will reach different parts of the airways and include; the mouth, the throat, the windpipe, and the bloodstream (all places we do not want the inhaled drug to go - and can give rise to important side effects)and, the lungs (where we do want the drug to 'deposit').

Our aim in this study is to test an inhaled steroid by giving it to subjects as a 'fine' mist containing drug particles of nearly all one size using a research nebuliser (a Spinning Top Aerosol Generator). We shall use small, intermediate and large drug particle mists. We aim to find out how much of the drug goes to the blood stream for each particle mist and compare it with the standard puffers used in routine clinical practice.

We hope this study will provide information to the rationale that by improving the efficiency of drug delivery (by changing drug particle size) one may improve inhaled drug delivery and ultimately, clinical patient benefit.

Healthy volunteers and asthmatic patients will be recruited at the Royal Brompton Hospital London. The study is funded by GlaxoSmithKline, Research & Development, U.K.

DETAILED DESCRIPTION:
The clinical trial is to investigate the pharmacokinetic effects (that is how much drug is in the blood) of Fluticasone Propionate (Flixotide), a commonly used steroid drug that is inhaled in patients with asthma. We will use standard clinical Flixotide Nebules that are used with clinical nebulisers (machines used in hospital and at home - to deliver drug to patients with asthma). Current clinical nebulisers deliver a 'coarse' mist of drug, which has the potential for side effects and this is an important consideration with steroids. These Flixotide nebules will be used to deliver the drug (fluticasone propionate) as monodisperse aerosol clouds (that is the drug will be delivered as a 'fine' mist cloud to patients). In order to deliver the drug as a monodisperse aerosol, the Flixotide Nebules will be used with a spinning top aerosol (a large research nebuliser machine)which is able to selectively generate aerosol clouds that have a fine mist. A fine mist cloud leads to less deposition in the throat of the patients and a greater control of the inhaled drug reaching the lungs, and fine mist drug clouds have the potential to reduce side effects. We will also compare this to the use of a standard routine clinical dose of a Flixotide metered-dose inhaler ( a 'press and breathe' inhaler) with a spacer (plastic bubble on the end of an inhaler) delivered to patients.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers

Participants will be included if they meet all of the following inclusion criteria

1. Healthy non smoking participants
2. Male or female aged above 18 years
3. No history of respiratory disease
4. Normal baseline spirometry as predicted for age, sex and height (we have excluded those with abnormal spirometry as this may indicate an underlying lung condition that needs attention, and such participants will be told their result and with their consent, the information will be forwarded to their General Practitioner, as part of the safety and well being of the research participant.
5. No history of allergic disease i.e., a negative skin prick test
6. Participants who are free from significant cardiac, gastrointestinal, hepatic, renal, hematological, neurological and psychiatric disease.
7. Not taking any regular medication that is contraindicated in those about to receive fluticasone propionate (as indicated in the British National Formularly); other than the oral contraceptive pill.

Asthmatics

1. Male or females aged greater than 18 years with a documented history of reversible airways disease responding to beta2-adrenergic therapy.
2. Asthmatic patients who are free from significant cardiac, gastrointestinal, hepatic, renal, hematological, neurological and psychiatric disease.
3. Patients who are stabilized on 500 micrograms or less of inhaled beclomethasone dipropionate or alternative inhaled corticosteroid (budesonide or ciclesonide).
4. Patients who are able and willing to give written informed consent to take part in the study
5. Not taking any regular medication that is contraindicated in those about to receive fluitcasone propionate (as indicated in the British National Formularly); other than the oral contraceptive pill.

Exclusion Criteria:

Healthy Volunteers and Asthmatics

1. Those requiring maintenance oral or parenteral corticosteroid therapy for their airways disease or patients who have ceased maintenance oral or parenteral corticosteroid therapy within the four weeks prior to visit 1
2. Those requiring greater than 500 micrograms of inhaled beclomethasone dipropionate or alternative inhaled corticosteroid (budesonide or ciclesonide).
3. Subjects that have received inhaled or intravenous fluticasone propionate in the last 2 months.
4. Those whose reversible airways obstruction has been unstable in the last four weeks (indicated by any change in their maintenance therapy).
5. Those participants who have had a lower respiratory tract infection in the previous four weeks
6. Those who have donated 450ml blood or more within the previous 1 month.
7. Those who have a history of drug allergy which, in the opinion of the Unit Physician, contraindicates his/her participation in the study.
8. Any evidence of a positive pregnancy urine test for female volunteers or females who are pregnant or lactating or are likely to become pregnant during the trial. Women of child-bearing potential may be included in the study if, in the opinion of the investigator, they are taking adequate contraceptive precautions.
9. Participants with a known or suspected allergy to corticosteroids or any component of the formulations and/or Suspected hypersensitivity to inhaled corticosteroid (this will be asked directly at the screening visit).
10. Any patient with a contraindication to taking an inhaled steroid and specifically FP, listed in the British National Formularly will not be entered into this study
11. Those who have experienced an acute asthma exacerbation requiring emergency room treatment and/or hospitalization within one month of visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2011-07-03 (Actual); Study Completion 2011-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: O S Usmani, MD, PhD, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Asthma Lab, Royal Brompton Hospital, London
  - Department of Nuclear Medicine, Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biddiscombe MF, Barnes PJ, Usmani OS. Generating monodisperse pharmacological aerosols using the spinning-top aerosol generator. J Aerosol Med. 2006 Fall;19(3):245-53. doi: 10.1089/jam.2006.19.245. PMID 17034300
- [Background] Usmani OS, Biddiscombe MF, Barnes PJ. Regional lung deposition and bronchodilator response as a function of beta2-agonist particle size. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1497-504. doi: 10.1164/rccm.200410-1414OC. Epub 2005 Sep 28. PMID 16192448
- [Background] Usmani OS, Biddiscombe MF, Nightingale JA, Underwood SR, Barnes PJ. Effects of bronchodilator particle size in asthmatic patients using monodisperse aerosols. J Appl Physiol (1985). 2003 Nov;95(5):2106-12. doi: 10.1152/japplphysiol.00525.2003. Epub 2003 Aug 1. PMID 12897033
- [Background] Biddiscombe MF, Usmani OS, Barnes PJ. A system for the production and delivery of monodisperse salbutamol aerosols to the lungs. Int J Pharm. 2003 Mar 26;254(2):243-53. doi: 10.1016/s0378-5173(03)00032-2. PMID 12623200

RESULTS

PARTICIPANT FLOW:
Groups:
- Asthma Patients; Healthy Volunteers: Monodisperse aerosols (MO) inhaled of Fluticasone Propionate (FP) 50micrograms dose
Period: FP From Active 250 ug MDI Inhaler
Arm/Group | Asthma Patients | Healthy Volunteers
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: FP1.5 Microns Size With MDI Inhaler
Arm/Group | Asthma Patients | Healthy Volunteers
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: FP 3 Microns Size With MDI Inhaler
Arm/Group | Asthma Patients | Healthy Volunteers
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: FP 6 Microns Size With MDI Inhaler
Arm/Group | Asthma Patients | Healthy Volunteers
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Asthma Patients: Recruited Asthma patients
- Healthy Volunteers: Recruited healthy volunteers
- Total: Total of all reporting groups
Arm/Group | Asthma Patients | Healthy Volunteers | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (11.8) | 35 (10.5) | 35 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 8 | 5 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: AUC Fluticasone Propionate (FP)
Description: The main outcome measure is the concentration of Fluticasone Propionate in blood following inhalation of the dose. This will be found by calculating the area under the curve of concentration versus time 0 and 12 hours.
Time Frame: 12 hours
Measure: Median (Full Range); unit: pg.h/ml
Groups:
- FP From Active 250 ug MDI Inhaler Asthma: Monodisperse aerosols inhaled of Fluticasone Propionate at 250micrograms dose with active MDI inhaler with Asthma participants
- FP 50ug 1.5um Asthma: Monodisperse aerosols inhaled of Fluticasone Propionate 1.5 microns size at 50micrograms dose with double-dummy placebo MDI inhaler with Asthma patients
- FP 50ug 3um Asthma: Monodisperse aerosols inhaled of Fluticasone Propionate 3 microns size at 50micrograms dose with double-dummy placebo MDI inhaler with Asthma patients
- FP 50ug 6um Asthma: Monodisperse aerosols inhaled of Fluticasone Propionate 6 microns size at 50micrograms dose with double-dummy placebo MDI inhaler with Asthma patients
- FP From Active 250 ug MDI Inhaler HV: Monodisperse aerosols inhaled of Fluticasone Propionate at 250micrograms dose with active MDI inhaler with Healthy participants
- FP 50ug 1.5um HV: Monodisperse aerosols inhaled of Fluticasone Propionate 1.5microns size at 50micrograms dose with double-dummy placebo MDI inhaler with Healthy volunteers
- FP 50ug 3um HV; FP 50ug 6um HV: Monodisperse aerosols inhaled of Fluticasone Propionate 3microns size at 50micrograms dose with double-dummy placebo MDI inhaler with Healthy volunteers
Arm/Group | FP From Active 250 ug MDI Inhaler Asthma | FP 50ug 1.5um Asthma | FP 50ug 3um Asthma | FP 50ug 6um Asthma | FP From Active 250 ug MDI Inhaler HV | FP 50ug 1.5um HV | FP 50ug 3um HV | FP 50ug 6um HV
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15
pg.h/ml | 188.2 [46.13 to 594.89] | 756 [613 to 2967] | 978 [413.8 to 2610.4] | 380.5 [2.2 to 1586.1] | 172.3 [34.4 to 778.41] | 740 [332 to 2421] | 934.6 [478 to 2647.7] | 250.4 [26.9 to 740.8]
Statistical Analysis 1: Comparison: FP From Active 250 ug MDI Inhaler Asthma vs FP 50ug 1.5um Asthma vs FP 50ug 3um Asthma vs FP 50ug 6um Asthma vs FP From Active 250 ug MDI Inhaler HV vs FP 50ug 1.5um HV vs FP 50ug 3um HV vs FP 50ug 6um HV; Test type: Equivalence — Log transformed parametric ANOVA; p < 0.05, ANOVA — calculated

ADVERSE EVENTS:
Time Frame: 4 months
Groups:
- FP From Active 250 ug MDI Inhaler Healthy: Monodisperse aerosols inhaled of Fluticasone Propionate at 250micrograms dose with active MDI inhaler with Healthy participants
- FP 50ug 1.5um Healthy: Monodisperse aerosols inhaled of Fluticasone Propionate 1.5 microns size at 50micrograms dose with double-dummy placebo MDI inhaler with Healthy participants
- FP 50ug 3um Healthy: Monodisperse aerosols inhaled of Fluticasone Propionate 3 microns size at 50micrograms dose with double-dummy placebo MDI inhaler with Healthy participants
- FP 50ug 6um Healthy: Monodisperse aerosols inhaled of Fluticasone Propionate 6 microns size at 50micrograms dose with double-dummy placebo MDI inhaler with Healthy participants
Arm/Group | FP From Active 250 ug MDI Inhaler Asthma | FP 50ug 1.5um Asthma | FP 50ug 3um Asthma | FP 50ug 6um Asthma | FP From Active 250 ug MDI Inhaler Healthy | FP 50ug 1.5um Healthy | FP 50ug 3um Healthy | FP 50ug 6um Healthy
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes